CLINICAL TRIAL: NCT03198195
Title: Post-transplant Cyclophosphamide for HLA-haploidentical Transplantation in Wiskott-Aldrich Syndrome
Brief Title: Post-transplant Cyclophosphamide in Wiskott-Aldrich Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Capital Research Institute of Pediatrics (Other Government)
Responsible Party: Principal Investigator, Yan Yue, MD,PhD, Capital Research Institute of Pediatrics
Other Study IDs: CIP-2015-08
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Wiskott-Aldrich Syndrome | interventions — Cyclophosphamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cyclophosphamide — on days +3，+4,using cyclophosphamide 50mg/kg

SUMMARY:
A protocol named as "CIP-2015" for patients with Wiskott-Aldrich Syndrome may reduce the rate of GvHD.

The details of the protocal followed with:

1. Conditioning regimen Busulfan 16 mg/kg in total, Fludarabine 160 mg/m2 in total.
2. GvHD Prophylaxis:

Rabbit antihuman thymocyte globulin 7.5 mg/kg post-transplant cyclophosphamide (CY) (50 mg/kg.d on days +3 and +4) Cyclosporine or tacrolimus, mycophenolate mofetil, on days +5

DETAILED DESCRIPTION:
Patients were enrolled in CIP-2015 Protocol at the Capital Institute of Pediatrics (Beijing). The conditioning regimen consisted of fludarabine (40 mg/m2) from days -6 to -3, and Busulfan was administered intravenously for 4 days, from days -5 to -2，using dose targeting based on therapeutic drug monitoring. Thymoglobulin (Sanoﬁ, Cambridge, MA) 7.5 to 10 mg/kg (cumulative dose over 4 days) was administered over 4 days, from days -5 to -2. Bone marrow (BM) and PBSC were infused on day 0, followed by post-transplant CY (50 mg/kg/day, on days +3 and +4). To protect against hemorrhagic cystitis, MESNA (2-mercaptoethane sodium sulfonate) was administered at 150% of the CY dose. Post grafting immunosuppression with mycophenolate mofetil and tacrolimus commenced on day +5 and extended until days +28 and +84, respectively. Tacrolimus was tapered off by day +90 if there was no GVHD.

ELIGIBILITY:
Inclusion Criteria:

-Patients diagnosed with Wiskott-Aldrich Syndrome with indication of Hematopoietic stem cell transplantation

Exclusion Criteria:

* without indication of Hematopoietic stem cell transplantation

Ages: 5 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient with Wiskott-Aldrich Syndrome :
  1. life-threatening bleeding
  2. strong demand of parents
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2020-07-10 (Estimated)

PRIMARY OUTCOMES:
Rate of aGvHD | 3month
  after post transplant cyclophospamide

IPD SHARING:
Plan to Share IPD: No